CLINICAL TRIAL: NCT03597893
Title: Effects of Intranasal Oxytocin and Induced Stress on People's Belief Updating
Brief Title: Effects of Intranasal Oxytocin and Stress on Belief Updating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OB-OT and stress
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: intranasal oxytocin; stress; belief updating
MeSH Terms: interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study utilized a randomized, double-blind, PBO controlled, between-subject design.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin (OXT), a neuropeptide produced in the hypothalamus, is a key modulator of complex socioaffective responses including affiliation, social approach and attachment, stress and anxiety. Subjects receiving an intranasal spray of OXT (24 IU or 40.32 mg; Syntocinon-spray; Novartis, Switzerland) .
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo contains all ingredients except for the peptide in three puffs of 3.99 IU per 6.72mg nostril.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasally administrated
  Arms: Oxytocin
Drug: Placebo — intranasally administrated
  Other Names: Saline
  Arms: Placebo

SUMMARY:
To investigate the effect of 24IU intranasal oxytocin on belief updating when people in stress or non-stress condition.

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo controlled between-subjects design, healthy male volunteers receive intranasal oxytocin or placebo under stress or non-stress group prior belief updating task.

The Trier Social Stress Test (TSST) was used to induce psychosocial stress - this standardized technique enables a naturalistic exposure to a psychosocially stressful situation. This method consists primarily of a public speaking in second language (English) and a mental arithmetic task performed in front of a panel. Participants were not informed of the tasks prior to their recruitment. At the start of the TSST, they were told to prepare a 5-min speech to an unknown panel on personal suitability for their ideal job; the job description was matched to each participant, taking into consideration his personal aspirations. After the instructions, subjects were given 10 minutes of solitary preparation for this task. Then, they entered the TSST room and were told to start the presentation in front of a panel of two formally-dressed judges (one male and one female) and a conspicuous video camera. Any pause during the speech prompted a reminder from the judges of the remaining time. The interview was followed by 5 minutes of mental arithmetic performed out loud. Subjects were instructed to serially subtract 13 from 1022 as quickly and accurately as possible in front of the panel. If a mistake was made, the subject was told to start over from the beginning. After the mental arithmetic task, the TSST was concluded - subjects were confronted with the psychosocially stressful situation for a total of 10 minutes.

Non-stress groups first underwent a 5-minute session of travel magazine reading with two casually-dressed people (one male and one female), then did as many easy arithmetic questions within 5 minutes on paper. Participants were told that none of their answers would be marked.

All participants completed two sessions of self life event estimations, each with the same set of 40 adverse life events. The subjects were first presented with the events, then were instructed to estimate their likelihood (0-99%) of experiencing each event in the future (first Estimate, E1) and rate their confidence in their estimate. They were then presented with the actual probability of each event occurring to an average person in a similar environment (Feedback, F) and asked to rate their acceptance of the presented feedback. Five minutes after the first session, participants were instructed to perform the same task and provide their second estimate (E2) for the same 40 events in a randomized order and were, again, instructed to rate their confidence in their estimate. This time, however, no feedback was given. This process was repeated for a friend life event estimation session. After the second session, participants were given a surprise memory test for the presented feedback.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* subjects with past or current psychiatric or neurological disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — we opted to recruit only males for the present study.
Enrollment: 131 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The updated probability estimation for negative events in the four experimental groups | 40~125 minutes after drug administration
  Using the second estimation value to minus the first estimation value to get the update value, as well as calculating the update value in desirable condition (first estimation < feedback) and undesirable condition (first estimation < feedback). Then investigated the general belief updating (gBU) and optimistic belief updating (using desirableBU-undesirableBU) in the four experimental condition (i.e., oxytocin-stress, oxytocin-nonstress, placebo-stress, placebo-nonstress).
The salivary cortisol level in four experimental groups | 40~125 minutes after drug administration
  Conducted ANOVA to test salivary cortisol level in the four experimental groups
The correlation between personality traits and belief updating value in four experimental groups | 40~125 minutes after drug administration
  Conducted correlation analysis to explore which personality traits would modulate the oxytocin effect or stress effect.